CLINICAL TRIAL: NCT04556773
Title: A Phase 1b Multicentre, Open-label, Modular, Dose-finding and Dose-expansion Study to Explore the Safety, Tolerability, Pharmacokinetics and Anti-tumour Activity of Trastuzumab Deruxtecan (T-DXd) in Combination With Other Anti-cancer Agents in Patients With Metastatic HER2-low Breast Cancer (DESTINY-Breast08)
Brief Title: A Phase 1b Study of T-DXd Combinations in HER2-low Advanced or Metastatic Breast Cancer
Acronym: DB-08
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Daiichi Sankyo Co., Ltd. (Industry); Daiichi Sankyo Company, Limited (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D967JC00002; 2023-505690-33-00 (Other: EU CT Number); 2020-002797-27 (EudraCT Number)
Record Dates: First submitted 2020-09-15; First posted 2020-09-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer; HER2-negative; HER2-low; Trastuzumab Deruxtecan; T-DXd; DS-8201a; DESTINY-Breast08; Anti-HER2 Antibody Drug Conjugate (ADC); Triple-negative breast cancer (TNBC)
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — trastuzumab deruxtecan; durvalumab; Paclitaxel; capivasertib; Anastrozole; Fulvestrant; Capecitabine

STUDY DESIGN:
Intervention Model Description: The study will initially consist of 5 treatment modules, each of which includes T-DXd in combination with other anti-cancer agents. Each module will have 2 parts: a dose-finding phase (Part 1) and a dose-expansion phase (Part 2). The Part 2 dose-expansion phase will use the recommended Phase 2 dose (RP2D) for the combination, either as determined in Part 1 or from another clinical study if appropriate. For each module, patients will be centrally assigned to one of the open modules, as per the module specific criteria.
  In addition to safety and tolerability, this study will also assess ORR, PFS, DoR, and OS for each treatment combination.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Module 1: T-DXd + capecitabine (Experimental): T-DXd: 5.4 mg/kg Q3W, intravenous use Capecitabine: 1000mg/m2 BID, days 1-14 Q3W, oral use
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Capecitabine
- Module 2: T-DXd + durvalumab + paclitaxel (Experimental): T-DXd: 5.4 mg/kg Q3W, intravenous use Durvalumab: 1120 mg Q3W, intravenous use Paclitaxel: 80 mg/m2 QW in 3-week cycles, intravenous use
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Durvalumab; Drug: Paclitaxel
- Module 3: T-DXd + capivasertib (Experimental): T-DXd: 5.4 mg/kg Q3W, intravenous use Capivasertib: 400 mg BID, oral use
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Capivasertib
- Module 4: T-DXd + anastrozole (Experimental): T-DXd: 5.4 mg/kg Q3W, intravenous use Anastrozole: 1 mg daily, oral
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Anastrozole
- Module 5: T-DXd + fulvestrant (Experimental): T-DXd: 5.4 mg/kg Q3W, intravenous use Fulvestrant: 500 mg Q4W, intramuscular use
  Interventions: Drug: Trastuzumab deruxtecan; Drug: Fulvestrant

INTERVENTIONS:
Drug: Trastuzumab deruxtecan — T-DXd: administered as an IV infusion
  Other Names: DS-8201a, T-DXd
Drug: Durvalumab — Durvalumab: administered as an IV infusion
  Other Names: MEDI4736
  Arms: Module 2: T-DXd + durvalumab + paclitaxel
Drug: Paclitaxel — Paclitaxel: administered as an IV infusion
  Other Names: Taxol A
  Arms: Module 2: T-DXd + durvalumab + paclitaxel
Drug: Capivasertib — Capivasertib: administered orally
  Other Names: AZD5363
  Arms: Module 3: T-DXd + capivasertib
Drug: Anastrozole — Anastrozole: administered orally
  Other Names: Anastrozol
  Arms: Module 4: T-DXd + anastrozole
Drug: Fulvestrant — Fulvestrant: administered as an IM injection
  Arms: Module 5: T-DXd + fulvestrant
Drug: Capecitabine — Capecitabine: administered orally
  Arms: Module 1: T-DXd + capecitabine

SUMMARY:
DESTINY-Breast 08 will investigate the safety, tolerability, PK and preliminary anti-tumour activity of T-DXd in combination with other therapies in patients with Metastatic HER2-low Advanced or Metastatic Breast Cancer

DETAILED DESCRIPTION:
This study is modular in design allowing assessment of the safety, tolerability, PK and preliminary anti-tumour activity of T-DXd in combination with other therapies. Combination-treatment modules will have 2 parts: a dose-finding phase (Part 1), and a dose expansion phase (Part 2); the Part 2 dose-expansion phase will use the RP2D determined in Part 1.

The target population of interest in this study is patients with HER2-low (IHC 1+ or IHC 2+/ISH -) (as per ASCO/CAP 2018 guidelines) advanced/MBC. Part 1 of each module will enroll patients with locally confirmed HER2-low advanced/MBC in second-line or later (≥ 2L) settings

Part 2 of each module will enroll patients with HER2-low MBC who have either not received prior treatment, or received only 1 prior treatment (depending on the module-specific exclusion criteria) for advanced/metastatic disease

ELIGIBILITY:
Key Inclusion Criteria:

* Patients must be at least 18 years of age
* Male or female patients who have pathologically documented breast cancer that:

  1. Has a history of HER2-low expression, defined as IHC 2+/ISH- or IHC 1+ (ISH- or untested) with a validated assay
  2. Is documented as HR+ (either ER and/or PgR positive [ER or PgR ≥1%]) or ER and PgR negative (ER and PgR <1%) per ASCO/CAP guidelines in the metastatic setting
* Patient must have adequate tumor sample for biomarker assessment
* ECOG Performance Status of 0 or 1

For patients with HR+ disease:

Part 1: At least 1 prior treatment line of ET with or without a targeted therapy (such as CDK4/6, mTOR or PI3-K inhibitors), and at least 1 prior line of chemotherapy for MBC are required.

Part 2: Only 1 prior treatment line of ET with or without a targeted therapy (such as CDK4/6, mTOR or PI3-K inhibitors) for MBC is allowed. No prior chemotherapy in the metastatic setting is allowed. Note there are no patients with HR+ disease in Part 2 of Modules 2 and 3.

For patients with HR- disease:

Part 1: At least 1 prior line of chemotherapy for MBC is required. Note there are no patients with HR- disease in Part 1 of Modules 4 and 5.

Part 2: For Module 2, no prior lines of therapy for MBC are allowed, and for Modules 1 and 3, only 1 prior line of chemotherapy for MBC is allowed. Note there are no patients with HR- disease in Part 2 of Modules 4 and 5.

Key Exclusion Criteria:

* Uncontrolled intercurrent illness
* Uncontrolled or siginificant cardiovascular disease
* History of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Lung-specific intercurrent clinically significant illnesses
* Has spinal cord compression or clinically active central nervous system metastases
* Active primary immunodeficiency
* Uncontrolled infection requiring IV antibiotics, antivirals, or antifungals
* Prior treatment with ADC that comprises of an exatecan derivative that is a topoisomerase I inhibitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2023-08-16 (Actual); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs)- Part 1 | Up to follow-up period, approximately 24 months
  Occurrence of AEs in Part 1 graded according to NCI CTCAE v5.0
Occurrence of serious adverse events (SAEs)- Part 1 | Up to follow-up period, approximately 24 months
  Occurrence of SAEs in Part 1 graded according to NCI CTCAE v5.0
Occurrence of adverse events (AEs)- Part 2 | Up to follow-up period, approximately 24 months
  Occurrence of AEs in Part 2 graded according to NCI CTCAE v5.0
Occurrence of serious adverse events (SAEs)- Part 2 | Up to follow-up period, approximately 24 months
  Occurrence of SAEs in Part 2 graded according to NCI CTCAE v5.0

SECONDARY OUTCOMES:
Objective Response Rate (ORR)- Part 2 | Until progression, assessed up to approximately 24 months
  ORR defined as the proportion of patients who have a confirmed CR or PR, as determined by the investigator at local site per RECIST 1.1
Progression Free Survival (PFS)- Part 2 | Until progression or death, assessed up to approximately 24 months
  PFS defined as time from the date of first dose until the date of progression as determined by the investigator at local site per RECIST 1.1, or death due to any cause
Duration of Response (DoR)- Part 2 | Until progression or death, assessed up to approximately 24 months
  DoR defined as time from the date of first documented response (which is subsequently confirmed) until the date of documented progression or death in the absence of disease progression
Overall Survival (OS)- Part 2 | Until death, assessed up to approximately 24 months
  OS defined as time from the date of first dose until the date of death by any cause
Serum concentration of T-DXd, total anti-HER2 antibody and MAAA-1181a | While on study drug up to study completion, approximately 24 months
  Determination of trastuzumab deruxtecan concentration in serum at different time points after trastuzumab deruxtecan administration
Immunogenicity of trastuzumab deruxtecan | Up to follow-up period, approximately 24 months
  Percentage of patients who develop ADA for trastuzumab deruxtecan
Serum Concentration of durvalumab | While on study drug up to study completion, approximately 24 months
  Determination of durvalumab concentration in serum at different time points after administration
Immunogenicity of durvalumab | Up to follow-up period, approximately 24 months
  Percentage of patients who develop ADAs for durvalumab

CONTACTS AND LOCATIONS:
Overall Officials: Komal Jhaveri, MD, FACP, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (27):
- United States (8):
  - Research Site, Commack, New York
  - Research Site, Harrison, New York
  - Research Site, New York, New York
  - Research Site, Uniondale, New York
  - Research Site, Chapel Hill, North Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Germantown, Tennessee
  - Research Site, Fort Worth, Texas
- Australia (2):
  - Research Site, East Melbourne
  - Research Site, Westmead
- Belgium (3):
  - Research Site, Edegem
  - Research Site, Leuven
  - Research Site, Ottignies
- Brazil (3):
  - Research Site, Goiânia
  - Research Site, Porto Alegre
  - Research Site, São Paulo
- Canada (2):
  - Research Site, Kelowna, British Columbia
  - Research Site, Québec, Quebec
- Research Site, Villejuif, France
- Research Site, Monterrey, Mexico
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- Research Site, Seoul, South Korea
- Taiwan (4):
  - Research Site, Kaohsiung City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: AstraZeneca Breast Cancer Study Locator website - To learn which AstraZeneca breast cancer clinical trials are looking for participants with specific diagnosis, stage, and treatment history. — http://BreastCancerStudyLocator.com
- See also: redacted Study Synopsis (core + module 1-5 (combined) — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D967JC00002&attachmentIdentifier=c690e364-5c63-4c87-b881-d6402fd48581&fileName=d967jc00002-study-synopsis-core,_module_1-5_(combined)_-_redacted.pdf&versionIdentifier=